CLINICAL TRIAL: NCT03376867
Title: Reference Values of Diffuse Noxious Inhibitory Controls (DNIC) Intensity in a Healthy Adult Population and Develop a Clinical Test to Evaluate DNIC
Brief Title: Reference Values and Clinical Screening Test of Diffuse Noxious Inhibitory Controls (DNIC)
Acronym: DNIC
Status: Active, not recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre for Research of CHUS (CRCHUS) (Unknown); CIHR/SPOR - chronic pain network (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-2422
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: conditioned pain modulation (CPM); Diffuse Noxious Inhibitory Controls (DNIC); pressure pain threshold (PPT); reference values; clinical decision rule
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be preserved as plasma (for biochemical analysis) and as Buffy coat cells (for genetic analysis on specific genes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Conditioned pain modulation (2 stimuli test: heat and pressure points) before and after conditioning stimuli (cold water bath).
  Interventions: Other: Conditioned pain modulation
- Volunteers with chronic pain: Conditioned pain modulation (2 stimuli test: heat and pressure points) before and after conditioning stimuli (cold water bath).
  Interventions: Other: Conditioned pain modulation

INTERVENTIONS:
Other: Conditioned pain modulation — Conditioned pain modulation (CPM) protocol consist of evaluating pain during two stimuli test (heat and pressure point), before and after one conditioning stimulus (cold water bath); Blood analyses for biochemistry and genes polymorphisms.
  Other Names: Pressure points

SUMMARY:
Chronic pain (CP) is disabling for people triggering important costs for society. A deficit of diffuse noxious inhibitory controls (DNIC) is one of the CP mechanisms. DNICs are evaluated in research setting using a CPM protocol (conditioned pain modulation). There is a lack of reference values on the effectiveness of DNICs. Wider research on DNIC will help to understand CP and to develop a clinical screening test evaluating DNICs.

DETAILED DESCRIPTION:
This study aims:

1. To establish baseline values of DNICs using CPM protocol
2. To identify the variables that will be integrated in the algorithm of the clinical screening test (clinical decision rule).

First the target population will be healthy volunteers, male and female, stratified by age. The reference values will be established via a non-parametric method for a standard CPM protocol in which two different pain stimuli are applied. Two "stimuli tests" of the same intensity and nature (heat) will be applied before and after the application of another "conditioning stimulus" (cold water bath). The perceived pain difference between the 1st and 2nd stimuli tests will reflect the intensity of the DNICs.

Secondly, these results will be compared to those from volunteers suffering of chronic pain. The clinical decision rule will result from clinical and paraclinical elements correlating with the amplitude of the efficacy of CPM (serum noradrenaline, intensity of pain, heart rate and blood pressure measurements, psychometric questionnaires assessing anxiety, depressive feelings and pain catastrophizing). Logistic regression analysis will determine the best predictors of a CPM deficit.

ELIGIBILITY:
Inclusion Criteria:

* 18-79 years old
* Able to provide consent

Exclusion Criteria:

* cardiovascular disease (arrhythmia, cerebrovascular accident, infarction...)
* Raynaud syndrome
* severe psychiatric disease (dementia, schizophrenia, psychosis, major depression)
* injuries or loss sensitivity to their forearms or hands
* pregnant women or in post-partum period (<1 year)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male and female volunteers (with no pain) will provide reference values to further study volunteers with chronic pain.
  People with chronic pain will constitute a second group to associate the conditioned pain modulation to their pain (chronic pain is defined by any regular pain for more than 6 months except pain caused by cancer or migraine)
Sampling Method: Probability Sample
Enrollment: 468 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Conditioned pain modulation | Once, at baseline, at recruitment (comparison between 1st and 2nd test, after the conditioning stimuli)
  Alteration (reduction or augmentation) of pain sensitivity after activation of endogenous pain-inhibitory system, measured by computerized visual analog scale (CoVAS) ranging from 0 [no pain] to 100 [most intense pain that could be tolerated]

SECONDARY OUTCOMES:
pressure points threshold | Twice, at baseline, at recruitment (before and after the conditioning stimuli)
  On both trapezius muscles

CONTACTS AND LOCATIONS:
Overall Officials: Louis Gendron, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Universite de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Vincenot M, Leonard G, Cloutier-Langevin C, Bordeleau M, Gendron L, Camirand Lemyre F, Marchand S. Exploring the Spectrum of Temporal Summation and Conditioned Pain Modulation Responses in Pain-Free Individuals Using a Tonic Heat Pain and Cold Pressor Test Paradigms. Eur J Pain. 2025 May;29(5):e70019. doi: 10.1002/ejp.70019. PMID 40176749